CLINICAL TRIAL: NCT02871557
Title: Frail Elderly Subjects Martinique: Adverse Outcome After Hospitalisation in Geriatric Department
Brief Title: Frailty and the Elderly in Martinique
Acronym: SAFMACohort
Status: Completed | Type: Observational
Sponsor: Société Martiniquaise de Gérontologie et Gériatrie (Other)
Collaborators: CHU de Reims (Other)
Responsible Party: Principal Investigator, Lidvine Godaert, Doctor, Société Martiniquaise de Gérontologie et Gériatrie
Other Study IDs: 1958830
Record Dates: First submitted 2016-08-11; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Elderly People With Polypathology or Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This was a prospective multicenter cohort study of elderly people admitted to the acute care for elders in Martinique. They were followed up to 36 months. It aimed to study the adverse outcomes. In all, 287 subjects were included. They were 85+/-6 years, and mainly women (61%).

DETAILED DESCRIPTION:
The SAFMA cohort was an ad hoc study formed into the recruitment of the acute care for elders in the geriatric department of Martinique university Hospitals. The inclusion of subjects ran from January 1st 2012 to June 30th 2012. To be eligible, patients had to be 75 or over and hospitalised for acute condition. Each patient was visited by a specialist in geriatrics familiar with the survey procedures. In the course of this interview, patients were informed about the study, prior to signing the consent form. If the clinical status and/or the cognitive status of the patient did not enable informed consent, the interviewer referred to the subject's representative. Follow-up was performed by visits and telephone interview till 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Age of 75 years or over
* Admitted to acute care for elders
* Consent to participate

Exclusion Criteria:

* Impossibility to perform the tests
* Refusals to participate

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A group of elderly people hospitalised in acute care for elders
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 weeks
Nursing home admission | 6 weeks

SECONDARY OUTCOMES:
Mortality | 6 month
Mortality | 12 month
Mortality | 24 month
Mortality | 36 month
Nursing home admission | 6 month
Nursing home admission | 12 month
Nursing home admission | 24 month
Nursing home admission | 36 month

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Godard-Sebillotte C, Drame M, Basileu T, Fanon JL, Godaert L. Is self-rated health an independent prognostic factor of six-week mortality in older patients hospitalized for an acute condition? Qual Life Res. 2016 Sep;25(9):2335-40. doi: 10.1007/s11136-016-1252-3. Epub 2016 Feb 26. PMID 26919847